CLINICAL TRIAL: NCT04802187
Title: Implementation of COVID-19 Testing Strategies in Community Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Harvard School of Public Health (HSPH) (Other); Massachusetts League of Community Health Centers (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elsie Taveras, MD, Executive Director, Kraft Center for Community Health and Division Chief, General Academic Pediatrics, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020P003743; 3P50CA244433-02S1 (NIH)
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Covid19
Keywords: implementation science; community health center
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RADx CHCs testing intervention strategy (Other): Six Massachusetts community health center partnerships implementing both a common testing expansion implementation strategy plus tailored strategies designed for community partner needs.
  Interventions: Other: RADx CHCs testing intervention strategy
- Usual care control (Other)
  Interventions: Other: Usual care control

INTERVENTIONS:
Other: RADx CHCs testing intervention strategy — The study team will support partner CHCs to implement workflows with some combination of dedicated testing staff, off-site testing, outreach/communications to priority populations, and linkage with local contact tracing systems. Implementation support will take the form of practice facilitation, rapid cycle testing (by supporting CHCs to review their internal data to assess the impact of workflow changes), and expert consultation from the research team on testing technology and testing location design.
  Arms: RADx CHCs testing intervention strategy
Other: Usual care control — CHCs implement testing strategies in accordance with their usual supports.
  Arms: Usual care control

SUMMARY:
This project is part of a competitive revision to accelerate COVID-19 testing in underserved populations. The overall aim is to implement strategies to expand COVID testing in hotspot communities in MA, through 6 community health center (CHC)-community partnerships. A base strategy will be implemented at all sites. A tailored strategy unique to local populations will be added and tested in a stepped wedge design.

ELIGIBILITY:
Inclusion Criteria:

* Participants are patients at the intervention or control CHCs or members of the local community. The participating sites constitute one group; a set of matched control CHCs that will conduct testing as usual constitute the second group.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elsie Taveras, MD, MPH, Principal Investigator — Massachusetts General Hospital; Karen Emmons, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Susan Dargon-Hart, LICSW, Principal Investigator — Massachusetts League of Community Health Centers
Locations (2):
- United States (2):
  - Massachusetts League of Community Health Centers, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled. 6 community health centers (CHC) contributed to control and intervention groups. These 6 CHCs were on the same time sequence in the interrupted time series and are listed as one group. To include an intervention and a control group separately would inaccurately sum the total participants to 12 CHCs. 6 CHCs contributed to both analytic groups (intervention and control). The study is therefore most accurately represented by including all CHCs in the same group.
Units Other Than Participants: Community health center
Groups:
- RADx CHCs Testing Intervention Strategy: Six Massachusetts community health center partnerships implementing both a common testing expansion implementation strategy plus tailored strategies designed for community partner needs.
  RADx CHCs testing intervention strategy: The study team will support partner CHCs to implement workflows with some combination of dedicated testing staff, off-site testing, outreach/communications to priority populations, and linkage with local contact tracing systems. Implementation support will take the form of practice facilitation, rapid cycle testing (by supporting CHCs to review their internal data to assess the impact of workflow changes), and expert consultation from the research team on testing technology and testing location design.
  All six community health centers had the same interruption point in the interrupted time series contributing 35 pre implementation usual care weeks, 85 post implementation intervention weeks.
Period: Overall Study
Arm/Group | RADx CHCs Testing Intervention Strategy
Started | NA; 6 Community health center (No participants were enrolled. 6 CHCs were in the primary analysis and completed the control and intervention milestones. Primary outcome was number of COVID tests. 186,171 Testing Intervention Strategy tests and 109,911 Usual Care tests collected.)
Completed | NA; 6 Community health center (No participants were enrolled. 6 CHCs were in the primary analysis and completed the control and intervention milestones. Primary outcome was number of COVID tests. 186,171 Testing Intervention Strategy tests and 109,911 Usual Care tests collected.)
Not Completed | NA; 0 Community health center

BASELINE CHARACTERISTICS:
Population: Participants were not enrolled into the study.
Units Other Than Participants: Number of tests
Groups:
- Total: Total of all reporting groups
Arm/Group | RADx CHCs Testing Intervention Strategy | Usual Care Control | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Number of tests) | 186171 | 109911 | 296082
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [19 to 51] | 38 [26 to 54] | 36 [22 to 52]
Sex/Gender, Customized [Count of Units; unit: Number of tests]
  Female | 107486 | 61507 | 168993
  Male | 78546 | 48322 | 126868
  Other | 47 | 40 | 87
  Unknown | 92 | 42 | 134
Ethnicity (NIH/OMB) [Count of Units; unit: Number of tests]
  Hispanic or Latino | 53751 | 28834 | 82585
  Not Hispanic or Latino | 107658 | 66222 | 173880
  Unknown or Not Reported | 24762 | 14855 | 39617
Race (NIH/OMB) [Count of Units; unit: Number of tests]
  American Indian or Alaska Native | 1094 | 512 | 1606
  Asian | 12662 | 5754 | 18416
  Native Hawaiian or Other Pacific Islander | 1923 | 994 | 2917
  Black or African American | 51987 | 25108 | 77095
  White | 69453 | 46358 | 115811
  More than one race | 229 | 0 | 229
  Unknown or Not Reported | 48823 | 31185 | 80008

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Testing During the Study Compared to Tests Completed Prior to Study Start
Description: Acceleration of covid testing volume during covid surges, estimated as the percent change in weekly covid testing volume trend for each 10% increase in covid cases. A slope value was estimated from a segmented regression model for the entire study period, which was then used to calculate a difference between the post- and pre-implementation periods.
Time Frame: 85 weeks post-implementation compared to 35 weeks pre-implementation
Population: No participants were enrolled in the study. The units analyzed represent the aggregate number of weekly COVID tests administered at the 6 community health centers.
Measure: Number (95% Confidence Interval); unit: Percent change
Units Other Than Participants: COVID tests
Groups:
- RADx CHCs Testing Intervention Strategy: Six Massachusetts community health center partnerships implementing both a common testing expansion implementation strategy plus tailored strategies designed for community partner needs for 85 weeks.
  RADx CHCs testing intervention strategy: The study team will support partner CHCs to implement workflows with some combination of dedicated testing staff, off-site testing, outreach/communications to priority populations, and linkage with local contact tracing systems. Implementation support will take the form of practice facilitation, rapid cycle testing (by supporting CHCs to review their internal data to assess the impact of workflow changes), and expert consultation from the research team on testing technology and testing location design.
- Usual Care Control: Usual care control: CHCs implement testing strategies in accordance with their usual supports for 35 pre implementation weeks.
Arm/Group | RADx CHCs Testing Intervention Strategy | Usual Care Control
Number analyzed (Participants) | NA | NA
Number analyzed (COVID tests) | 186171 | 109911
Percent change | 0.0965 [.04 to .153] | 0.0128 [-0.003 to 0.028]

ADVERSE EVENTS:
Description: Patients were not recruited for the intervention. Enrolled study participants were community health centers. Therefore adverse event reporting did not apply.
Arm/Group | RADx CHCs Testing Intervention Strategy | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT04802187/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT04802187/SAP_001.pdf